CLINICAL TRIAL: NCT03159884
Title: The Efficacy Assessment of Intravitreal Injection of Conbercept in Patients With Polypoidal Choroidal Vasculopathy (PCV)
Acronym: STAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KH902-ST-CRP-2.0
Record Dates: First submitted 2017-02-08; First posted 2017-05-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-02

CONDITIONS: Polypoidal Choroidal Vasculopathy (PCV)
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — KH902 fusion protein

ARMS (2):
- 3+Q12W (Experimental): The eye of interest will first receive three consecutive intravitreal injections of 0.5 mg conbercept every 4 weeks, followed by every 12 weeks. If the subject meets the "additional medication criteria" in 12 weeks during treatment, additional injection can be given;
  Interventions: Drug: Conbercept
- 3+TAE (Experimental): The eye of interest will first receive three consecutive intravitreal injections of 0.5 mg conbercept every 4 weeks, then the researcher will determine the next follow-up visit time/treatment interval based on results of each follow-up assessment as per the "treatment-extended dosing criteria". When the follow-up/treatment interval of the subject is extended to 12 weeks, additional safety follow-up visit can be arranged if any suspicious active lesion is deemed by the researcher; additional injection can be given if the result of safety follow-up assessment meets the "extra dosing criteria".
  Interventions: Drug: Conbercept

INTERVENTIONS:
Drug: Conbercept

SUMMARY:
To assess the efficacy of intravitreal injection of 0.5 mg conbercept in patients with polypoidal choroidal vasculopathy (PCV) and explore the optimal route of administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has signed an informed consent form and is inclined to be followed up within the time stipulated in the trial;
* Patient with wet AMD aged ≥ 45, of either sex;
* The eye of interest must meet the following requirements:

  1. BCVA is at least 19 and at most 83 alphabets (equivalent to a visual acuity of 20/25 to 20/400 for the Snellen Eye Chart);
  2. Patient has been diagnosed with active PCV on ICGA (confirmed by the third-party radiodiagnosis center); The diagnostic criteria for "active" PCV on ICGA are as follows: image indicates polypoid lesions as typical nodular high fluorescein area (observed stereoscopically) and also depicts one of the following angiographic findings: 1) nodular lesions surrounded by the weak halo; 2) nodular lesions nourished by abnormal vascular beds; and 3) nodular pulsation on dynamic ICGA;
  3. In case of the eye of interest complicated with subretinal hemorrhage or hemorrhage under the pigment epithelium, the range of hemorrhage should not be beyond the upper and lower vascular arcades in the macular area, and the total thickness of the central fovea (i.e., the thickness between the apex of the central fovea and the choriocapillary layer) is no more than 600 µm;
  4. Neither ocular media opacity nor miosis is noted to influence the fundus examination.
* Subject with the BCVA of no less than 19 alphabets for his/her eye of non-interest (equivalent to a visual acuity of 20/400 for the Snellen Eye Chart).

Note: Each subject in the study can include only one eye of interest; the eye of interest is determined by the researcher from a medical point of view if both eyes of the subject meet the inclusion criteria.

Exclusion Criteria:

* Subfoveal fibrous tissues are present in the eye of interest on CFP and OCT;
* Researcher judges that existing or previous ocular diseases in the eye of interest influence the macular detection or the central visual acuity (CNV secondary to diseases other than AMD, diabetic retinopathy, uveitis, angioid streaks, pathologic myopia, retinal pigment epithelium (RPE) tears, macular holes, any retinal vasculopathy, vein occlusion, amblyopia, retinal inflammatory diseases, central serous choroidopathy, previous or existing retinal detachment, macular edema, anterior ischemic optic neuropathy, pseudovitelliform macular degeneration, vitreomacular traction syndrome, rhegmatogenous retinal detachment, generalized choroidal atrophy, and optic atrophy (pale));
* There is any history of vitreous hemorrhage three months before screening;
* The eye of interest has received any drug therapy for AMD (e.g., pegaptanib sodium or steroids) or any anti-VEGF therapy (e.g., ranibizumab or bevacizumab);
* The eye of interest has received verteporfin-photodynamic therapy (PDT) and foveal laser-induced thermal therapy (including subfoveal or paracentral photocoagulation, grid photocoagulation, transpupillary thermotherapy (TTT) and pan-retinal photocoagulation);
* The eye of interest has received intra- or periocular surgery (including parafoveal laser photocoagulation treatment, cataract surgery, and YAG laser posterior capsulotomy) within three months, except eyelid surgery having no effect on intravitreal injection (but eyelid surgery could not be performed one month before medication);
* The eye of interest has received the following ophthalmic operations, including vitrectomy, macular translocation, glaucoma surgery, laser photocoagulation and pan-retinal photocoagulation, as well as other submacular surgeries or other surgeries for CNV;
* The eye of interest has received keratoplasty;
* Either eye has active eye infection (e.g., blepharitis, infective conjunctivitis, keratitis, scleritis, and endophthalmitis) or recurrent infection, or the eye of interest has been infected 30 days before screening;
* Patient has either previous or existing uncontrollable glaucoma (defined as IOP remaining at above 25 mmHg after anti-glaucoma treatment), or the cup-to-disc ratio of the eye of interest is above 0.8 due to severe glaucoma, or the eye of interest has received glaucoma filtration surgery;
* No ruptured lens (excluding pseudophakic) or posterior lens capsule (except YAG laser posterior capsulotomy after intraocular lens implantation);
* Patient needs to receive cataract surgery three months after enrollment (i.e., the researcher judges that BCVA may decrease by no less than 10 alphabets for the subject if the surgery is not performed);
* The eye of interest has ocular tumor;
* There is a history of systemic use of anti-VEGF agent(s) in six months;
* Patient has a history of anaphylaxis and allergy to fluorescein sodium and indocyanine green, and of allergy to protein products for diagnosis or treatment, and is allergic to no less than two drugs and/or non-drug factors, or suffers from allergic diseases now;
* Diabetics with uncontrolled blood glucose (fasting blood glucose ≥ 7.0 mmol/L or 2hPBG ≥ 11.1 mmol/L) and/or complicated with diabetic retinopathy;
* Patient has had a surgical history one month before enrollment, and/or has unhealed wounds, ulcers and fractures at present;
* Patient has infectious diseases required oral, intramuscular or intravenous administration at present;
* Patient has a history of myocardial and/or cerebral infarction(s) within 6 months before screening, has received stenting and depends on such anticoagulants as warfarin and aspirin;
* Patient chronically uses and cannot discontinue to use such anticoagulants as aspirin, clopidogrel and warfarin;
* Patient has active and disseminated intravascular coagulation and distinct bleeding tendency three months before screening;
* Hyperpietics with poor blood pressure control (defined as blood pressure remaining at ≥ 150/95 mmHg after antihypertensives therapy);
* Patient is diagnosed with systemic immune disease (e.g., ankylosing spondylitis, systemic lupus erythematosus, and Behcet's disease) or has any uncontrollable clinical problem (e.g., AIDS, malignancies, active hepatitis, renal failure, severe mental, neurological, cardiovascular and respiratory diseases);
* Patient has previously used drugs which may possibly cause renal toxicity, including chloroquine, hydroxychloroquine, phenothiazines, chlorpromazine, thioridazine, fluphenazine, perphenazine, and trifluoperazine;
* Patient does not take effective contraceptive measures; Note: The following conditions are not included in the exclusion range.

  1. Amenorrhea for 12 months under the natural condition, or amenorrhea for 6 months under the natural condition and the serum FSH level of > 40 mIU/ml;
  2. Six weeks after bilateral ovariectomy with/without hysterectomy;
  3. Use of the following one or more acceptable contraceptions:

     * Sterilization (for males, with bilateral vasoligation and vasectomy)
     * Hormonal contraception (implantable, patchable, oral)
     * Intrauterine device and dural barrier method
  4. Ability to take reliable contraceptive measures over the study period and hold on to 30 days after study drug withdrawal (unacceptable contraceptive methods include: periodic continence - according to the calendar and ovulatory phase, body thermometry, post-ovulatory method, and coitus interruptus).
* Pregnant women (in this trial pregnancy is defined as positive U-HCG) and breastfeeding mothers;
* Patient has participated in any drug (not including vitamins and minerals) clinical trial three months before screening (if the study drug has a long half-life, i.e., its five half-lives exceed three months, then it is deemed as five half-lives); Those whom the reseacher deems necessary to exclude.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change of Best Corrected Visual Acuity | Baseline, 12th and 48th week
  The investigators will use the ETARS Chart which is international standard to measure the vision ability of participants.Best corrected visual is the number of letters which the participants can read on the ETARS Chart ,all procedure should be done according to SOP.The BCVA of 12th week and 48th week will be compared with the base line（pre-treatment）.

SECONDARY OUTCOMES:
Central Retinal Thickness (CRT) | week 48
  To observe pre- and posttreatment changes in CRT on OCT
Change of Macular Retinal Thickness (MRT) | week 48
  To observe pre-and posttreatment changes on OCT;
Volume and Thickness of Retinal Pigment Epithelial Detachment (PED) | week 48
  To observe pre- and posttreatment changes in volume and thickness of PED on OCT;
Area and Regression of Polypoidal Lesion | week 48
  To observe pre- and posttreatment changes in area and regression of polypoidal lesion on ICGA
Size of Retinal Hemorrhages | week 48
  To observe pre- and posttreatment changes in size of retinal hemorrhages on CFP
Area of Branching Vascular Network | week 48
  To observe pre- and posttreatment changes in area of BVN on ICGA
Frequency of Administration | up to 48 weeks
  Refers to the average frequency of administration for both groups of subjects during the study.
Incidence of adverse events (AEs) and reactions | up to 48 weeks
Ophthalmic examination | up to 48 weeks
  Ophthalmic examination include corneal、vitreous body、anterior chamber、iris、retina、disc、Macular 、drusen、PED examination Investigator will check whether the parts above is normal. Measurement for summarizing the data : Number of patients with different conditions of each part.
General symptoms and vital signs | up to 48 weeks
  Number of participants with abnormal symptoms or vital signs.
Number of participants with adverse events as assessed by laboratory results | up to 48 weeks
  Laboratory results include Blood routine 、Blood biochemistry、Coagulation function 、Urine routine 、Urinary pregnancy .
Number of participants with treatment-related adverse events as assessed by other tests. | up to 48 weeks.
  Other tests indicated that which is not contained in the study done by the participants .

CONTACTS AND LOCATIONS:
Locations (35):
- China (35):
  - Beijing Hospital, Beijing
  - Beijing Shijitan Hoospital.Cmu, Beijing
  - Beijing Tongren Hospital,Cmu, Beijing
  - Chinese Pla General Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People'S Hospital, Beijing
  - PEKING UNIVERSITY Third HOSPITAL, Beijing
  - The Scond Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital Central South University, Changsha
  - General Hospial og Guangzhou Military Command of PLA, Guangzhou
  - ZhongShan Ophthalmic Center,Sun Yat-sen University, Guangzhou
  - Hainan Eye Hospital of Zhongshan Ophthalmic Center, Sun Yat-sen University, Hainan
  - Hebei Eye Hospital, Hebei
  - The Second Hospital of Hebei Medical University, Hebei
  - Henan Province People's Hospital, Henan
  - The Second Hospital of Jilin University, Jilin
  - Lanzhou University Second Hospital, Lanzhou
  - Affiliated Eye Hospital of Nanchang University, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing General Hospital, Nanjing
  - The First Affiliated Hospital With Nanjing Medical University, Nanjing
  - Ningxia Peple'S Hospital, Ningxia
  - Eye&Ent Hospital of Fudan University, Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Stu/Cuhk Joint Shantou International Eye Center, Shantou
  - Shanxi Eye Hospital, Shanxi
  - Shenzhen Eye Hospital, Shenzhen
  - Tianjin Medical University Eye Hospital, Tianjin
  - The Chinese people's liberation army 474 hospital, Ürümqi
  - The Eye Hospital of Wmu Zhejiang Eye Hospital, Wenzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - Xiamen Eye Centre of Xiamen University, Xiamen
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Zhejiang